CLINICAL TRIAL: NCT07151807
Title: Evaluation of Serum IGF-1 and IGF-1Ec (E-peptide/MGF) Levels and Their Association With Tumor Burden in Patients With Solid Tumors
Brief Title: Serum IGF-1 and IGF-1Ec in Malignancy Assessment
Acronym: SIGMA
Status: Active, not recruiting | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Cemre Aydeğer, Research asistant, PhD, Çanakkale Onsekiz Mart University
Other Study IDs: COMU-FNO-4
Record Dates: First submitted 2025-07-31; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Solid Tumor Malignancies; IGF1R; Solid Cancers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: The study group will consist of at least 60 adult patients (aged 18 and older) with histologically confirmed solid tumors who are clinically stable and have not yet started or are in the early phase of standard chemotherapy. Participants will be recruited from the outpatient and inpatient oncology units at Çanakkale Onsekiz Mart University. Individuals with hematological malignancies, organ failure, or conditions/medications affecting IGF-1 levels will be excluded.

SUMMARY:
This cross-sectional study investigates the relationship between serum IGF-1 and IGF-1Ec (E-peptide/MGF) levels and tumor burden in patients with solid tumors. By analyzing serum samples using ELISA and correlating them with clinical data such as tumor stage, size, metastasis, and lymph node involvement, the study aims to explore whether these biomarkers-particularly IGF-1Ec and the IGF-1Ec/IGF-1 ratio-can reflect tumor progression and serve as potential prognostic indicators.

DETAILED DESCRIPTION:
Background: Insulin-like Growth Factor-1 (IGF-1) and its splice variant IGF-1Ec (also known as Mechano Growth Factor, MGF) play critical roles in cell proliferation, survival, and tumor progression. Recent evidence suggests that IGF-1Ec may act independently of the classical IGF-1 receptor pathway and contribute to aggressive tumor behavior. However, data on serum IGF-1Ec levels and their correlation with clinical tumor burden remain limited.

Objective: This cross-sectional analytical study aims to quantify serum IGF-1 and IGF-1Ec levels in patients with solid tumors and investigate their association with tumor burden parameters such as clinical stage, tumor size, lymph node involvement, and metastasis. The IGF-1Ec/IGF-1 ratio will also be evaluated as a potential prognostic biomarker.

Methods: Serum samples will be collected from approximately 60 patients diagnosed with solid tumors. IGF-1 and IGF-1Ec levels will be measured using validated ELISA kits. Clinical tumor burden will be assessed from medical records (TNM staging, metastasis, tumor diameter). Statistical analysis will include group comparisons and correlation tests.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed diagnosis of a solid tumor
* Clinically stable condition, prior to chemotherapy or during standard follow-up
* Ability to provide informed consent

Exclusion Criteria:

* Hematological malignancies (e.g., leukemia, lymphoma)
* Acute or chronic liver or kidney failure
* Current use (within 1 month) of corticosteroids, growth hormone, or medications affecting IGF-1 levels
* Pregnancy or lactation
* Coagulopathy or severe anemia preventing safe venipuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include approximately 100 adult patients (≥18 years old) diagnosed with histologically confirmed solid tumors. All participants will be recruited from the Çanakkale Onsekiz Mart University Oncology Outpatient Clinic or Inpatient Services. Only clinically stable patients will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
IGF-1 and IGF-1Ec levels | From enrollment to 6 month
  Blood values

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided